CLINICAL TRIAL: NCT01660646
Title: A Cluster Randomised Trial to Assess the Impact of an Enhanced Case Finding Strategy on Tuberculosis Notification in The Gambia
Brief Title: Determining the Impact of Enhanced Case Finding on Tuberculosis Notification in The Gambia
Acronym: ECF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SCC 1205
Record Dates: First submitted 2012-07-26; First posted 2012-08-09 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Tuberculosis
Keywords: Tuberculosis case finding
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral: community sensitization (Other): Behavioral, enhanced case finding (ECF) by community sensitization via audiovisual presentation in local languages, a session for questions and answers and opportunity to provide sputum specimens for detection of TB
  Interventions: Behavioral: Behavioral: community sensitization
- control (No Intervention)

INTERVENTIONS:
Behavioral: Behavioral: community sensitization — Behavioral, enhanced case finding (ECF) by community sensitization via audiovisual presentation in local languages, a session for questions and answers and opportunity to provide sputum specimens for detection of TB
  Arms: Behavioral: community sensitization

SUMMARY:
This is a cluster Tuberculosis (TB) randomized trial in which enhanced case finding (ECF) strategy will be compared to passive TB case reporting in The Gambia. And that the impact of ECF on community and household transmission of TB will also be assessed.

The hypothesis is a cluster randomized trial of an enhanced case finding (ECF) strategy will increase TB case notifications in The Gambia and reduce TB burden in the study area in a cost effective manner. The impact of ECF on community and household transmission of TB will also be assessed. The investigators hope this trial will contribute to this evidence base. The timing alongside a nationwide TB prevalence survey is particularly of benefit as that would provide a baseline for disease burden against which the investigators may be able to compare case notification or case detection in selected clusters

DETAILED DESCRIPTION:
TB is a chronic, transmissible disease, albeit with effective and curative combination therapeutic regimens available. However insufficient case detection, delayed diagnosis of TB , which prolong the duration of potential transmission, and co prevalent HIV/AIDS are the major factors responsible for increasing TB incidence. The DOTs strategy, which relies on a process of passive TB case finding, has helped to control TB in many parts of the world. Currently, the World Health Organisation's Stop TB DOTS policy is being questioned as countries that have reached and maintained targets of 70% case detection and 85% cure rates are unable to demonstrate a decline in number of cases notified.

Studies in Southern Africa suggest that if the investigators want to prevent TB in HIV-infected and uninfected people a major focus should be on decreasing transmission from people who are HIV-negative that may transmit TB for a long time on account of delayed diagnosis 5, 6. Data from studies in Ethiopia, Peru, Brazil, and Zimbabwe show different strategies of intensified or active case finding (ICF or ACF) yield significantly more TB cases than the standard of care-passive case finding.7-10 In the Zimbabwe study, point prevalence of TB declined significantly over 2 time points and was attributed to the ICF intervention. Since effective treatment for TB renders patients non-infectious within 2-4 weeks, it is likely that earlier diagnosis and initiation of treatment will ultimately reduce the incidence of TB by interrupting TB transmission. However the quantitative effect of enhanced case finding (ECF) on TB case notification rates, TB transmission, prevalence and incidence remains largely unproven.

Although there is now data from Zimbabwe regarding the impact of untargeted active case finding strategies, it is unclear how each case finding strategy compares to the standard passive case finding and the investigators are currently unable to address the cost effectiveness or otherwise of active case finding strategies in high TB burden settings with low HIV prevalence which is the scenario in most West African countries including The Gambia. Consequently, there is insufficient data to support a policy change and an urgent need for evidence to drive the necessary review of policy.

The hypothesis is a cluster randomized trial of an enhanced case finding (ECF) strategy will increase TB case notifications in The Gambia and reduce TB burden in the study area in a cost effective manner. The impact of ECF on community and household transmission of TB will also be assessed. The investigators hope this trial will contribute to this evidence base. The timing alongside a nationwide TB prevalence survey is particularly of benefit as that would provide a baseline for disease burden against which the investigators may be able to compare case notification or case detection in selected clusters.

ELIGIBILITY:
Inclusion Criteria:

* Any newly diagnosed case initiating TB therapy at any of the Gambia Government TB diagnostic and treatment centres in the Greater Banjul Area.
* All TB patients are eligible regardless of age, residency, HIV status, or type of TB
* All settlements randomised to the intervention arm

Exclusion Criteria:

* Inability to understand the implications of study participation, whether through cognitive impairment or insurmountable language barrier.
* Communities that refuse to accept intervention through decision conveyed by the alkalo and other recognised community leaders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 650000 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The total number of successive TB cases notified in the intervention area compared to the total number of successive TB cases notified in the control areas | 30 months

SECONDARY OUTCOMES:
The total cost of making diagnosis and receiving treatment will be compared between ECF and passive case finding | 30 months
  Residual burden of TB after intervention Proportion of TB detected through ECF vs. passive case finding in intervention areas.
  Evaluation of diagnostic delay and treatment outcome in cases detected through ECF versus passive case finding

CONTACTS AND LOCATIONS:
Overall Officials: Ifedayo Adetifa, FWACP, MSc, Principal Investigator — Medical Research Council Unit, The Gambia
Locations (1):
- Medical Research Council Unit, The Gambia, Fajara, Near Banjul, The Gambia